CLINICAL TRIAL: NCT05866952
Title: Quantitative Computed Tomography to Assess Ventilatory and Perfusion Abnormalities in Individuals With Post-Acute Sequelae of SARS-CoV-2 Infection
Brief Title: Ventilatory and Perfusion Abnormalities in Individuals With Post-Acute Sequelae of SARS-CoV-2 Infection
Acronym: PASC VQ
Status: Recruiting | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: 4DMedical (Industry)
Responsible Party: Sponsor
Other Study IDs: 2337
Record Dates: First submitted 2023-05-16; First posted 2023-05-19 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Post-Acute COVID-19; Post COVID-19 Condition; Post Viral Fatigue; Dyspnea
Keywords: Ventilation Perfusion Mismatch
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Post-Acute Sequelae of SARS-CoV-2 (PASC) Group: Subjects with PASC with a documented history of COVID-19 and persistent symptoms of fatigue, dyspnea, and/or exercise intolerance
  Interventions: Diagnostic Test: Computed Tomography of the Chest
- Control: Fully recovered COVID-19: Subjects with a history of COVID-19 who have fully recovered from COVID-19 with no post-acute sequelae of SARS-Cov-2
  Interventions: Diagnostic Test: Computed Tomography of the Chest
- Control: No history of COVID-19: Healthy subjects without a documented history of COVID-19, no current symptoms, and a normal baseline High resolution CT of the chest
  Interventions: Diagnostic Test: Computed Tomography of the Chest

INTERVENTIONS:
Diagnostic Test: Computed Tomography of the Chest — Quantitative Computed Tomography of the chest in the inspiratory and expiratory phases will be performed to assess regional lung ventilation as well as pulmonary vascular volume and distribution

SUMMARY:
Prospective cohort study to evaluate the utility of quantitative CT analysis to assess ventilation and perfusion defects in patients with Post-acute Sequelae of SARS-CoV-2 (PASC) and functional limitations

DETAILED DESCRIPTION:
This is a study to describe the overall pattern of lung ventilation and perfusion defects in individuals with PASC. Subjects with PASC with a documented history of COVID-19 and persistent symptoms of fatigue, dyspnea, and/or exercise intolerance will complete questionnaires, and undergo pulmonary function tests, 6-minute walk tests, and a low dose CT chest to describe the overall pattern of lung regional ventilation and blood distribution and to compare this pattern to asymptomatic controls with and without prior COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Self-reported or documented SARS-CoV-2 infection by RT-PCR or Antigen testing > 3 months ago or no previous history of SARS-CoV-2 infection (control group only)
* Normal or mild abnormalities on baseline Pulmonary Function Tests (PFTs)
* New or worsening symptoms of chronic fatigue, dyspnea or exercise intolerance after COVID-19 with otherwise unclear etiology (PASC group only)

Exclusion Criteria:

* SARS-CoV-2 infection by RT-PCR or Antigen testing within the last 3 months
* Inability to provide consent or non-English speaking
* Pregnancy
* Any respiratory infection in last 4 weeks
* PFT relative contraindications
* History of major cardiovascular, pulmonary, renal, hepatic, autoimmune or neuromuscular disease including asthma, COPD, interstitial lung disease, heart failure, pulmonary arterial hypertension, or prior pulmonary embolism
* Active malignancy undergoing treatment or history of malignancy involving the lung

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The primary population of interest includes participants with a history of COVID-19 who continue to have symptoms of dyspnea, fatigue, or exercise intolerance 3 months beyond their initial infection. The comparison cohorts will include 2 controls: individuals fully recovered from prior COVID-19 and healthy controls without a history of COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measures of regional lung ventilation | 1 day
Measures of blood volume distribution | 1 day

SECONDARY OUTCOMES:
Dyspnea severity scores | 1 day
Fatigue severity scores | 1 day
Quality of life scores | 1 day
Six-minute walk distance | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States